CLINICAL TRIAL: NCT05075174
Title: Effect of Progesterone Levels on 15th Day After Embryo Transfer in Early Miscarriage < 7 WG or Evolving Pregancy Rates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0564
Record Dates: First submitted 2021-09-18; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: ART
Keywords: betaHCG +; pregnancy development know; progesterone level; miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Progesterone level has been studied at days before embryo transfert. But, progesterone blood level has not been studied 15 days after embryo transfert. The aim of this study is to study progesterone level impact at 15 days after embryo transfert on evolving pregnanies or early miscarriages.

ELIGIBILITY:
Inclusion criteria:

* ART program in Montpellier hospital
* age >18 years old
* Blood progesterone level 15 days after embryo transfert
* Pregnancy development know

Exclusion criteria:

- non uterine pregnancy

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: ART program in Montpellier hospital >18 years old Blood progesterone level 15 days after embryo transfert Pregnancy development know
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
number of blood progesterone | 1 day
  blood progesterone at day 15 after embryo transfert

CONTACTS AND LOCATIONS:
Overall Officials: Noémie Ranisavljevic, M.D., Ph.D, Study Director — University Hospital, Montpellier; MARIE DUPORT PERCIER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC